CLINICAL TRIAL: NCT02421679
Title: A 12-Week, Open-Label, Multicenter, Extension Study To TNX-CY-P201 To Evaluate The Safety And Efficacy Of TNX-102 SL Taken Daily At Bedtime In Patients With Military-Related PTSD And Related Conditions
Brief Title: Open Label Extension Safety and Efficacy Study of TNX-102 SL Tablets in Military Related PTSD and Related Conditions
Acronym: P202
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNX-CY-P202
Record Dates: First submitted 2015-04-09; First posted 2015-04-21 (Estimated); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: PTSD
Keywords: PTSD; Military-related PTSD and other related conditions; open-label extension
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TNX-102 SL (Experimental): TNX-102 SL taken daily at bedtime for 12 weeks
  Interventions: Drug: TNX-102 SL

INTERVENTIONS:
Drug: TNX-102 SL — 1x 2.8mg TNX-102 SL Sublingual tablet
  Other Names: cyclobenzaprine HCI

SUMMARY:
This is a 12-week, multicenter, open-label extension study to evaluate the safety and efficacy of TNX-102 SL tablet taken daily at bedtime in patients with Military-Related PTSD or related condition. Patients recruited into this trial are those who have successfully completed the double-blind study, TNX-CY-P201 (AtEase Study) [NCT02277704]. Patients will not be made aware of the therapy they received during the double-blind study.

DETAILED DESCRIPTION:
The study will consist of 4 clinic visits, including Screening/Baseline Visit 1 (Day 0, which is anticipated to be the same date as the final visit in the lead-in P201 study) and visits after 2, 6 and 12 weeks of treatment. The previous requirements in the lead-in study for refraining from the use of certain concomitant medications and trauma-focused psychotherapies will be relaxed. Patients may continue to take rescue therapy for sleep, as appropriate, or they may utilize other medications as needed to help them sleep, per the judgment of the investigator.

Eligible patients who provide written informed consent will take one TNX-102 SL tablet daily at bedtime sublingually (under the tongue) for 12 weeks. All patients will be assigned to receive tthe same dosage of TNX-102 SL, regardless of their treatment assignment in the lead-in study. No patients, investigators, or study staff will know the assigned study treatment from the lead-in study, P201, at the time of entry into the extension study. Patient data collected at the Week 12 visit (Visit 9) in the lead-in P201 study will be used as one of the baseline values for this study.

ELIGIBILITY:
Inclusion Criteria:

* Completed the lead-in study and is judged as reasonably compliant, with at least 60% compliance
* Signed informed consent
* Met all prior inclusion and exclusion requirements for lead-in study
* No new or worsening medical conditions since starting the lead-in study that could pose a safety risk or interfere with participation in the study
* Willing to refrain from use of specific medication (ask PI)
* Female patients of childbearing potential continue to practice medically acceptable methods of birth control

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2016-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Bedoya, Study Director — Premier Research
Locations (22):
- United States (22):
  - Tuscaloosa VA Medical Center, Tuscaloosa, Alabama
  - Noesis Pharma, Phoenix, Arizona
  - Sun Valley Research Center, Imperial, California
  - Synergy Clinical Research, National City, California
  - Excell Research, Inc, Oceanside, California
  - Neuropsychiatric Research Center of Orange County, Orange, California
  - CITRIALS, Riverside, California
  - CESAMH, San Diego, California
  - Cns, Inc., Torrance, California
  - Sarkis Clinical Trials, Lake City, Florida
  - Compass Research North, LLC, Leesburg, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Atlanta Center For Medical Research, Atlanta, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Novex Clinical Research, New Bedford, Massachusetts
  - Premier Psychiatric Research Institute, Inc., Lincoln, Nebraska
  - Altea Research, Las Vegas, Nevada
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Clinical Trials of Texas, San Antonio, Texas
  - Northwest Clinical Research Center, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo- TNX-102 SL 2.8 mg: These patients received 2x Placebo sublingual tablets daily at bedtime during the lead-in study (TNX-CY-P201) and 1x TNX-102 SL 2.8 mg tablet daily at bedtime during this open-label study.
- TNX 102 SL 2.8 mg - TNX-102 SL 2.8 mg: These patients received 1x TNX-102 SL 2.8 mg sublingual tablet and 1x Placebo sublingual tablet daily at bedtime during the lead-in study (TNX-CY-P201) and 1x TNX-102 SL 2.8 mg tablet daily at bedtime during this open-label study.
- TNX-102 SL 5.6 mg - TNX-102 SL 2.8 mg: These patients received 2x TNX-102 SL 2.8 mg sublingual tablets daily at bedtime during the lead-in study (TNX-CY-P201) and 1x TNX-102 SL 2.8 mg tablet daily at bedtime during this open-label study.
Period: Overall Study
Arm/Group | Placebo- TNX-102 SL 2.8 mg | TNX 102 SL 2.8 mg - TNX-102 SL 2.8 mg | TNX-102 SL 5.6 mg - TNX-102 SL 2.8 mg
Started | 58 | 64 | 37
Completed | 47 | 49 | 32
Not Completed | 11 | 15 | 5

BASELINE CHARACTERISTICS:
Population: Numbers are only reported for the safety population, which includes all patients who received at least one dose of investigational product under this protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo- TNX-102 SL 2.8 mg | TNX 102 SL 2.8 mg - TNX-102 SL 2.8 mg | TNX-102 SL 5.6 mg - TNX-102 SL 2.8 mg | Total
Number analyzed (Participants) | 54 | 60 | 35 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (7.00) | 35.8 (8.22) | 35.4 (9.27) | 34.7 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 10
  Male | 50 | 57 | 32 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 8 | 5 | 24
  Not Hispanic or Latino | 43 | 52 | 30 | 125
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 3 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 16 | 8 | 33
  White | 36 | 41 | 25 | 102
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 4 | 1 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 54 | 60 | 35 | 149

OUTCOME MEASURES:

1. Primary Outcome: Newly Treatment Emergent Adverse Events
Description: Number of patients with new treatment emergent AEs since completing lead-in study
Time Frame: Week 12
Population: Results are reported for the safety population, which includes all patients who received at least one dose of investigational product under this protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo- TNX-102 SL 2.8 mg | TNX 102 SL 2.8 mg - TNX-102 SL 2.8 mg | TNX-102 SL 5.6 mg - TNX-102 SL 2.8 mg
Number analyzed (Participants) | 54 | 60 | 35
Participants | 37 | 20 | 14

2. Secondary Outcome: Total CAPS-5 (Clinician Administered PTSD Scale (for Diagnostic and Statistical Manual of Mental Disorders Version 5)
Description: Changes in total CAPS-5 score from baseline in lead-in study and since baseline in this study. CAPS-5 score ranges from 0-80 with lower scores indicating less sever PTSD symptoms.
Time Frame: P201 Day 1 (12 weeks prior to P202 Day 1), P202 Day 1, P202 Week 12
Population: Only patients with data available at all timepoints were evaluated.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo- TNX-102 SL 2.8 mg | TNX 102 SL 2.8 mg - TNX-102 SL 2.8 mg | TNX-102 SL 5.6 mg - TNX-102 SL 2.8 mg
Number analyzed (Participants) | 48 | 51 | 33
units on a scale
  Change from P201 Baseline to P202 Week 12 | -25.3 (2.55) | -25.6 (2.59) | -26.9 (2.80)
  Change from P202 Baseline to P202 Week 12 | -4.9 (1.80) | -4.8 (1.82) | -3.7 (2.01)

3. Secondary Outcome: Response Rates a in Total CAPS-5 Score
Description: ≥30% decrease in Total CAPS-5 score from baseline in lead-in study and since baseline in this study. Lower scores on CAPS-5 indicate less severe PTSD symptoms.
Time Frame: P201 Day 1 (12 weeks prior to P202 Day 1), P202 Day 1, P201 Week 12
Population: Any patients with missing values are assigned as not achieving 30% improvement.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo- TNX-102 SL 2.8 mg | TNX 102 SL 2.8 mg - TNX-102 SL 2.8 mg | TNX-102 SL 5.6 mg - TNX-102 SL 2.8 mg
Number analyzed (Participants) | 54 | 60 | 35
Participants
  Patients with ≥30% decrease in Total CAPS-5 score from P201 Day 1 to P202 Week 12 | 43 | 47 | 30
  Patients with ≥30% decrease in Total CAPS-5 score from P202 Day 1 to P202 Week 12 | 20 | 24 | 13

4. Secondary Outcome: CAPS-5 Cluster Score Items
Description: Changes from baseline in lead-in study and since baseline in this study in item scores, including
  * intrusion symptoms (Criterion B) - Score ranges from 0 to 20.
  * CAPS-5 item 2. (B-2) (unpleasant dreams related to the trauma) - Score ranges from 0 to 4
  * persistent avoidance (Criterion C) - Score ranges from 0 to 8
  * negative cognitions and mood (Criterion D) - Score ranges from 0 to 28
  * arousal and reactivity (Criterion E) - Score ranges from 0 to 24 Lower scores indicate less severe symptoms on all items
Time Frame: P201 Day 1 (12 weeks prior to P202 Day 1), P202 Day 1, P202 Week 12
Population: Only patients with data available at all timepoints were evaluated.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo- TNX-102 SL 2.8 mg | TNX 102 SL 2.8 mg - TNX-102 SL 2.8 mg | TNX-102 SL 5.6 mg - TNX-102 SL 2.8 mg
Number analyzed (Participants) | 48 | 51 | 33
units on a scale
  Change from P201 Day 1 to P202 Week 12 in Criterion B | -7.7 (0.82) | -7.4 (0.82) | -7.7 (0.91)
  Change from P202 Day 1 to P202 Week 12 in Criterion B | -1.9 (0.66) | -1.5 (0.66) | -1.4 (0.74)
  Change from P201 Day 1 to P202 Week 12 in Item B-2 | -1.3 (0.23) | -1.4 (0.24) | -1.4 (0.26)
  Change from P202 Day 1 to P202 Week 12 in Item B-2 | -0.3 (0.20) | -0.4 (0.21) | -0.2 (0.23)
  Change from P201 Day 1 to P202 Week 12 in Criterion C | -3.1 (0.45) | -3.2 (0.45) | -3.1 (0.50)
  Change from P202 Day 1 to P202 Week 12 in Criterion C | -0.4 (0.38) | -0.5 (0.39) | -0.5 (0.42)
  Change from P201 Day 1 to P202 Week 12 in Criterion D | -7.6 (1.10) | -8.4 (1.12) | -9.1 (1.22)
  Change from P202 Day 1 to P202 Week 12 in Criterion D | -1.1 (0.85) | -1.8 (0.85) | -1.4 (0.95)
  Change from P201 Day 1 to P202 Week 12 in Criterion E | -6.8 (0.83) | -6.4 (0.84) | -7.1 (0.91)
  Change from P202 Day 1 to P202 Week 12 in Criterion E | -1.4 (0.62) | -0.9 (0.62) | -0.8 (0.69)

5. Secondary Outcome: Montgomery-Asberg Depression Rating Scale
Description: Changes from baseline in lead-in study and since baseline in this study in MADRS. Score ranges from 0 to 60. Lower scores indicate less severe depression symptoms.
Time Frame: P201 Day 1 (12 weeks prior to P202 Day 1), P202 Day 1, P202 Week 12
Population: Only patients with data available at all timepoints were evaluated.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo- TNX-102 SL 2.8 mg | TNX 102 SL 2.8 mg - TNX-102 SL 2.8 mg | TNX-102 SL 5.6 mg - TNX-102 SL 2.8 mg
Number analyzed (Participants) | 48 | 51 | 33
units on a scale
  Change from P201 Day 1 to P202 Week 12 | -8.1 (1.53) | -9.3 (1.57) | -9.9 (1.66)
  Change from P202 Day 1 to P202 Week 12 | 0.1 (1.28) | -1.1 (1.30) | -2.1 (1.40)

6. Secondary Outcome: PROMIS (Patient -Reported Outcome Measurement Information System)
Description: Changes from baseline in lead-in study and since baseline in this study in PROMIS scores. Raw scores are converted to T-scores with mean of 50 and standard deviation of 10 using published conversion tables based on the US population.
  * Fatigue T-score ranges from 33.1 to 77.8. Lower scores indicate less fatigue
  * Sleep Disturbance T-score ranges from 28.9 to 76.5. Lower scores indicate less sleep disturbance
  * Global Physical Health T-score ranges from 16.2 to 67.7. Lower scores indicate better physical health
  * Global Mental Health T-score ranges from 21.2 to 67.6. Lower scores indicate better mental health
Time Frame: P201 Day 1 (12 weeks prior to P202 Day 1), P202 Day 1, P202 Week 12
Population: Only patients with data available at all timepoints were evaluated.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo- TNX-102 SL 2.8 mg | TNX 102 SL 2.8 mg - TNX-102 SL 2.8 mg | TNX-102 SL 5.6 mg - TNX-102 SL 2.8 mg
Number analyzed (Participants) | 48 | 51 | 32
T-score
  Change from P201 Day 1 to P202 Week 12 in PROMIS Sleep Disturbance T-scores | -10.4 (2.50) | -12.2 (2.58) | -14.3 (2.75)
  Change from P202 Day 1 to P202 Week 12 in PROMIS Sleep Disturbance T-scores | 0.7 (2.36) | 0.4 (2.40) | -3.1 (2.60)
  Change from P201 Day 1 to P202 Week 12 in PROMIS Fatigue T-scores | -5.6 (2.05) | -6.4 (2.08) | -8.0 (2.26)
  Change from P202 Day 1 to P202 Week 12 in PROMIS Fatigue T-scores | 0.9 (1.78) | 1.1 (1.79) | -0.4 (1.93)
  Change from P201 Day 1 to P202 Week 12 in PROMIS Global Mental Health T-scores | 7.1 (1.76) | 7.1 (1.79) | 10.1 (1.95)
  Change from P202 Day 1 to P202 Week 12 in PROMIS Global Mental Health T-scores | 0.5 (1.50) | 0.2 (1.53) | 1.8 (1.67)
  Change from P201 Day 1 to P202 Week 12 in PROMIS Global Physical Health T-scores | 3.1 (1.50) | 3.2 (1.53) | 5.8 (1.66)
  Change from P202 Day 1 to P202 Week 12 in PROMIS Global Physical Health T-scores | -0.7 (1.18) | -0.2 (1.20) | 1.7 (1.30)

ADVERSE EVENTS:
Time Frame: 12 Weeks
Description: All adverse events are reported for the Safety population, which includes only the patients who took at least 1 dose of study medication in this study.
Arm/Group | Placebo- TNX-102 SL 2.8 mg | TNX 102 SL 2.8 mg - TNX-102 SL 2.8 mg | TNX-102 SL 5.6 mg - TNX-102 SL 2.8 mg
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/60 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/60 | 0/35
Other Adverse Events (participants affected / at risk) | 29/54 | 7/60 | 3/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo- TNX-102 SL 2.8 mg (N=54) | TNX 102 SL 2.8 mg - TNX-102 SL 2.8 mg (N=60) | TNX-102 SL 5.6 mg - TNX-102 SL 2.8 mg (N=35)
Hypoaesthesia Oral (Gastrointestinal disorders) | 22 | 3 | 2
Paraesthesia Oral (Gastrointestinal disorders) | 9 | 1 | 0
Somnolence (Nervous system disorders) | 2 | 3 | 1
Product Taste Abnormal (Product Issues) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA is in place with all investigators.